CLINICAL TRIAL: NCT01242462
Title: Feasibility of Mid-frequency Ventilation in Newborn Infants With Respiratory Distress Syndrome (RDS): Crossover Pilot Trial
Brief Title: Feasibility of Mid-frequency Ventilation in Newborns With RDS: Randomized Crossover Pilot Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ramachandra Bhat, MD, Fellow Instructor, Department of Pediatrics, Division of Neonatology, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UAB NEO 002
Record Dates: First submitted 2010-11-15; First posted 2010-11-17 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: Conventional mechanical ventilation; Mid-frequency ventilation; Respiratory Distress Syndrome; Preterm Newborn Infant; Mean Airway Pressure; Mean Arterial Pressure; Mean Peak Inspiratory Pressure
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AB (Active Comparator): 2 hours of treatment with conventional ventilation strategy, then crossover to 2 hours of treatment with mid-frequency ventilation strategy
  Interventions: Procedure: Conventional Pressure Controlled SIMV; Other: Mid-frequency Ventilation
- BA (Active Comparator): 2 hours of treatment with mid-frequency ventilation strategy, then crossover to 2 hours of treatment with conventional ventilation strategy
  Interventions: Procedure: Conventional Pressure Controlled SIMV; Other: Mid-frequency Ventilation

INTERVENTIONS:
Procedure: Conventional Pressure Controlled SIMV — Initial ventilatory settings per clinical physician's discretion-tcCO2 & Saturation (SAT) monitoring. Adjust vent setting approximately every 15min with a goal of: SAT 88-95%, tcCO2 45-55, pH greater than or equal to 7.25. Once goals reached, ventilatory strategy will crossed over to other intervention.
Other: Mid-frequency Ventilation — Ventilatory parameters include: max possible rate between 61-150 breaths/min; Shortest inspiration time (Ti) and expiration time (Te), but completed inspiration and expiration on pulmonary graphics. Stepwise weaning of PIP by 1 cm H20 to maintain tcCO2 at baseline. If measured PEEP - delivered PEEP generated is >/= to 1cm H2O, PEEP is reduced to baseline value. Adjustments will be made to PIP, then rate for pH and CO2 changes; FiO2, then PIP for FiO2 changes. Target goal blood gas parameters (same as baseline) Saturations 88-95%; tcCO2 45-55 mmHG; pH >/= 7.25. Maximum period of 2 hours. When goals met, or 2 hours in period, reverted back to SIMV at baseline settings

SUMMARY:
Respiratory distress syndrome (RDS) is the most common respiratory disorder in preterm infants. Despite improved survival of extremely premature infants with RDS, complications related to mechanical ventilation still occur. This trial will attempt to maintain adequate gas exchange at a rapid rate, short inspiratory time, low tidal volume, and low peak inspiratory pressure in infants with respiratory distress requiring mechanical ventilation. A cross over design will be used to test the hypothesis whether mid-frequency ventilation in preterm infants with RDS requiring mechanical ventilation will reduce the peak inspiratory pressure requirement when compared to conventional mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Inborn newborn infants with birthweight greater than or equal to 500gms, with gestational age greater than or equal to 24 weeks but less than or equal to 36 weeks.
* Postnatal age less than or equal to 7 days.
* Infant with respiratory distress syndrome (RDS) on mechanical ventilation with less than or equal to 60 breaths/minute, initially requiring greater than or equal to 30% FiO2.
* Written informed consent.

Exclusion Criteria:

* Blood culture positive sepsis, life threatening congenital anomalies, cyanotic congenital heart diseases, hydrops fetalis, outborn infants, non viability as determined by the attending physician, and newborns who are considered too unstable for study enrollment as per neonatology attending/fellow.

Ages: 1 Hour to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Average delta pressure | 4 hours
  Difference in peak inspiratory pressure (PIP) and peak end expiratory pressure (PEEP) (average delta pressure) during two time periods--time period on conventional synchronized intermittent ventilation (SIMV) and time period on mid-frequency ventilation, randomly assigned.

SECONDARY OUTCOMES:
Average Mean Airway Pressure (MAP) | Less than 4 hours
  Comparison of mean airway pressure between 2 periods of ventilation--(A)Conventional ventilation strategy and (B)Mid-frequency ventilation
Mean arterial pressure | Less than 4 hours
  Comparison of mean arterial pressure during two periods of mechanical ventilation--(A)Conventional ventilation strategy and (B)Mid-frequency ventilation
Average delta pressure | Less than 4 hours
  Comparison of average delta pressure during the two periods of mechanical ventilation-(A)Conventional ventilation strategy and (B)Mid-frequency ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Ramanchandra Bhat, MD, Principal Investigator — University of Alabama at Birmingham; Waldemar A Carlo, MD, Study Director — University of Alabama at Birmingham; John Kelleher, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Bhat R, Kelleher J, Ambalavanan N, Chatburn RL, Mireles-Cabodevila E, Carlo WA. Feasibility of Mid-Frequency Ventilation Among Infants With Respiratory Distress Syndrome. Respir Care. 2017 Apr;62(4):481-488. doi: 10.4187/respcare.05157. Epub 2017 Jan 3. PMID 28049742